CLINICAL TRIAL: NCT04500236
Title: Release of Serum Neurofilament Light (NFL), Biomarker of Neuronal Injury, in Surgery Under General Anaesthesia (GA) Compared to Surgery With Hypno-analgesia (Hyp): A Prospective, Non-inferiority Study
Brief Title: Serum Neurofilament Light (NFL) in Surgery Under General Anaesthesia (GA) Compared to Surgery With Hypno-analgesia (Hyp)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/14MAI/273
Record Dates: First submitted 2020-07-22; First posted 2020-08-05 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: General Surgery
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (GA) (Active Comparator): Patients undergoing thyroid or breast cancer surgery under general anesthesia
  Interventions: Other: General anesthesia
- Hypno-analgesia (Hyp) (Placebo Comparator): Patients undergoing thyroid or breast cancer surgery under Hypno-analgesia; i.e.hypnosis combined with the use of analgesics.
  Interventions: Other: Hypno-analgesia

INTERVENTIONS:
Other: General anesthesia — Surgery under general anesthesia with the use of propofol
  Arms: General Anesthesia (GA)
Other: Hypno-analgesia — Surgery under Hypnosis session and analgesics
  Arms: Hypno-analgesia (Hyp)

SUMMARY:
Experimental studies have shown that inhalational anesthetics may be neurotoxic by for example causing amyloid beta deposition. Otherwise a pre-clinical study reported an increase in tau phosphorylation with the use of propofol.

Whether anesthesia and surgery contribute to the development of long-term cognitive decline remains however controversial. A meta-analysis concluded that general anesthesia could increase the risk of postoperative cognitive decline (POCD) compared with regional or combined anesthesia but this was not shown for Postoperative delirium (POD). This conclusion should be interpreted with caution as these studies showed many shortcomings.

Currently no study has compared the release of Neurofilament Light, a biomarker of neuronal injury, in patients undergoing surgery under general anesthesia compared to surgery with Hypno-analgesia and thus without anesthetic drugs.

DETAILED DESCRIPTION:
POD and POCD are manifestations of cognitive dysfunction occurring in the perioperative period. Whether surgery and specifically anesthesia contribute to the development of perioperative cognitive dysfunctions is not clear.

Cell culture and animal studies have suggested detrimental effects of anesthetic exposure.1,2,3 Otherwise, it has been shown in animals that surgery plus anesthesia produced worse POCD than anesthesia alone.4 Proinflammatory cytokine levels increase during surgery. These elevated levels of inflammatory markers associated with the activation of microglial cells may induce neuroinflammation enhancing ongoing neurodegeneration.5 However, anesthetics may be capable of modulating inflammation and may alter the neuroinflammatory response.

Clinical studies associating the effects of general anesthesia with POCD and POD are conflicting.6 These varying results could be due to heterogeneity of patients' baseline status (e.g. cognitive status, education, associated diseases), type of surgery, as well as methods used to determine POCD and POD.

The use of serum neurobiomarkers, sensitive and specific for neuronal cell injury will address the hypothesis of general anesthesia neurotoxicity. Serum Neurofilament Light (NFL) is such a neurobiomarker.Currently no study has compared the release of Neurofilament Light, a biomarker of neuronal injury, in patients undergoing surgery under general anesthesia compared to surgery with Hypno-analgesia and thus without anesthetic drugs. Our hypothesis is that surgery under GA compared to hypnosis does not statistically increase the risk of neuronal injury as measured by serum NFL.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing thyroid or breast cancer surgery and necessitating one night of hospital stay

Exclusion Criteria:

* Renal insufficiency with a GFR < 30 mL/min
* Mammectomy
* Preoperative psychiatric problems
* Patients not speaking fluently French
* Patients at risk of postoperative hyperalgesia (Kalkman score > 4/15)
* Allergy to local anesthetics, NSAID and to Rocuronium
* Patients undergoing one day surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Serum Neurofilament Light at first postoperative day (18 - 24 hours) postoperatively) between both groups | 18 hours to 24 hours postoperatively
  Comparison of postoperative serum Neurofilament Light between both groups

SECONDARY OUTCOMES:
Total postoperative analgesic consumption between both groups | 24 hours postoperatively
  Comparison of total consumed analgesics in the postoperative period
Postoperative C-reactive protein between both groups | 24 hours postoperatively
  Comparison of postoperative highest C-reactive protein between both groups
Postoperative serum Neurofilament Light in function of type of surgery | 24 hours postoperatively
  Analysis of postoperative serum Neurofilament Light in function of type of surgery
Comparison of postoperative Montreal Cognitive Assessment on a scale of 30 (higher scores are better) between both groups | Day 8 to day 10
  Postoperative Montreal Cognitive Assessment
Postoperative serum Neurofilament Light at postoperative day 8 - 10 | Day 8 to day 10
  Analysis of postoperative serum Neurofilament Light between both groups
Quality of Recovery F15 questionnaire with 15 questions on a scale of 10 (higher scores are better) between both groups | Day 8 to day 10
  Comparison of quality of recovery between both groups based on a validated questionnaire with 15 items

OTHER OUTCOMES:
Frontal EEG analysis of patients under hypnosis | Intraoperatively
  Analysis of raw frontal EEG power (in slow, delta, theta, alpha, beta and gamma band) from the depth-of-anesthesia monitor as a sub-analysis of this study

CONTACTS AND LOCATIONS:
Overall Officials: Mona Momeni, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
All data will be available at the moment of publication of results

REFERENCES:
- [Background] Whittington RA, Virag L, Marcouiller F, Papon MA, El Khoury NB, Julien C, Morin F, Emala CW, Planel E. Propofol directly increases tau phosphorylation. PLoS One. 2011 Jan 31;6(1):e16648. doi: 10.1371/journal.pone.0016648. PMID 21304998
- [Background] Eckenhoff RG, Johansson JS, Wei H, Carnini A, Kang B, Wei W, Pidikiti R, Keller JM, Eckenhoff MF. Inhaled anesthetic enhancement of amyloid-beta oligomerization and cytotoxicity. Anesthesiology. 2004 Sep;101(3):703-9. doi: 10.1097/00000542-200409000-00019. PMID 15329595
- [Background] Wei H, Xie Z. Anesthesia, calcium homeostasis and Alzheimer's disease. Curr Alzheimer Res. 2009 Feb;6(1):30-5. doi: 10.2174/156720509787313934. PMID 19199872
- [Background] Wan Y, Xu J, Ma D, Zeng Y, Cibelli M, Maze M. Postoperative impairment of cognitive function in rats: a possible role for cytokine-mediated inflammation in the hippocampus. Anesthesiology. 2007 Mar;106(3):436-43. doi: 10.1097/00000542-200703000-00007. PMID 17325501
- [Background] Riedel B, Browne K, Silbert B. Cerebral protection: inflammation, endothelial dysfunction, and postoperative cognitive dysfunction. Curr Opin Anaesthesiol. 2014 Feb;27(1):89-97. doi: 10.1097/ACO.0000000000000032. PMID 24300462
- [Background] Mason SE, Noel-Storr A, Ritchie CW. The impact of general and regional anesthesia on the incidence of post-operative cognitive dysfunction and post-operative delirium: a systematic review with meta-analysis. J Alzheimers Dis. 2010;22 Suppl 3:67-79. doi: 10.3233/JAD-2010-101086. PMID 20858956